CLINICAL TRIAL: NCT01687374
Title: Phase IV Study of the Effect of Parathyroid Hormone on Fractures of the Humerus
Brief Title: Parathyroid Hormone for the Treatment of Humerus Fractures
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, Ulrich Bang, Principal investigator, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HvH-2011-545-1
Record Dates: First submitted 2012-03-12; First posted 2012-09-18 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Shoulder Fractures
Keywords: proximal humeral fracture
MeSH Terms: conditions — Shoulder Fractures | interventions — Parathyroid Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Parathyroid hormone (Experimental)
  Interventions: Drug: 1-84 parathyroid hormone

INTERVENTIONS:
Drug: 1-84 parathyroid hormone — 100 micrograms of 1-84 parathyroid hormone daily for 8 weeks, subcutaneous injection.
  Arms: Parathyroid hormone
Drug: Placebo — Saline injection daily for 8 weeks.
  Arms: Placebo

SUMMARY:
Hypothesis:

The investigators want to study whether parathyroid hormone improves healing of humerus after a fracture. The investigators will assess healing of the humerus with Constant score.

ELIGIBILITY:
Inclusion Criteria:

* proximal humeral fracture eligible for conservative treatment.
* able to understand the protocol
* signs an informed consent

Exclusion Criteria:

* liver disease
* kidney disease
* severe osteoporosis
* malignant disease
* bone metabolic disease
* oral treatment with bisphosphonates during the last 3 months.
* treatment with Denosumab during the last 6 months.
* intravenous treatment with bisphosphonates during the last 12 months.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Changes in constant score | 5, 8, 11, 23, and 104 weeks.
  Constant score summarizes the function of the arm using a questionnaire (activities of daily living - ADL) and functional testing of the arm.

SECONDARY OUTCOMES:
Changes in Oxford Shoulder Score | 5, 8, 11, 23, and 104 weeks.
  Oxford shoulder score is a questionnaire that assesses the function of the arm through the evaluation of the participant.
Changes in bone formation evaluated by X-ray. | 5, 8, 11, 23, and 104 weeks.
Changes in biochemical bone markers | 0, 5, 25 weeks
  sodium, potassium, creatinine, liver enzymes, vitamin D, parathyroid hormone, alkaline phosphatase, hemoglobin, magnesium, calcium, zinc.
Changes in regulatory T lymphocytes | 0, 8, 24 weeks
  Regulatory CD3+CD4+CD25+Foxp3+ T lymphocytes.

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre Hospital, Hvidovre, Denmark

REFERENCES:
- [Background] Aspenberg P, Genant HK, Johansson T, Nino AJ, See K, Krohn K, Garcia-Hernandez PA, Recknor CP, Einhorn TA, Dalsky GP, Mitlak BH, Fierlinger A, Lakshmanan MC. Teriparatide for acceleration of fracture repair in humans: a prospective, randomized, double-blind study of 102 postmenopausal women with distal radial fractures. J Bone Miner Res. 2010 Feb;25(2):404-14. doi: 10.1359/jbmr.090731. PMID 19594305
- [Background] Peichl P, Holzer LA, Maier R, Holzer G. Parathyroid hormone 1-84 accelerates fracture-healing in pubic bones of elderly osteoporotic women. J Bone Joint Surg Am. 2011 Sep 7;93(17):1583-7. doi: 10.2106/JBJS.J.01379. PMID 21915572